CLINICAL TRIAL: NCT00740974
Title: Allergy and Asthma Following Children Who Were Fed Supplemented Infant Formula
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Other Study IDs: 8580
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Allergy; Asthma
MeSH Terms: conditions — Hypersensitivity; Asthma

SUMMARY:
Long-term cognitive outcome study of children who participated in randomized trials of LCP-supplemented formula during infancy.

ELIGIBILITY:
Inclusion Criteria:

* children previously randomized in a clinical study consuming LCP-supplemented infant formula

Exclusion Criteria:

* children who did not previously participate in a randomized clinical study consuming LCP-supplemented infant formula

Ages: 5 Days to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children previously randomized in a clinical study consuming LCP-supplemented infant formula

PRIMARY OUTCOMES:
Prevalence of asthma and allergy related diagnosis in medical records during first 3 years of life. | after first 3 years of life

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Foundation of the Southwest, Dallas, Texas, United States